CLINICAL TRIAL: NCT05668650
Title: Randomized, Multicenter, Multinational, Double-blind Study to Evaluate the PK, Efficacy, Safety and Immunogenicity of MB12 (Proposed Pembrolizumab Biosimilar) Versus Keytruda® in Subjects With Stage IV NSCLC
Brief Title: Double-blind Study to Evaluate the PK, Efficacy, Safety and Immunogenicity of MB12 Versus Keytruda® in Stage IV NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB12-C-01-22
Record Dates: First submitted 2022-12-12; First posted 2022-12-30 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Non Small Cell Lung Cancer Metastatic
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a randomized, multicenter, multinational, double-blind, and parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be double-blind during the whole study period. The double-blind design reduces the potential for bias, particularly in the assessment of AEs. Most of the other assessments in the current study are objective in nature and, therefore, less prone to bias.
  The blinding for a specific subject can be broken by the investigator (emergency code breaking) only if the investigator considers the information indispensable to the safety of the subject. All subjects whose treatment are unblinded by the investigator (break blind option, emergency code breaking) while on the study will be withdrawn at the moment of unblinding, with the reason for unblinding given as the reason for discontinuation from the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Reference Product (Active Comparator): Keytruda® will be administered as monotherapy, on Day 1 of every 3-week cycle (21 days), during the Main Study Period (6 cycles) unless there is disease progression, intolerance to the study drug, or treatment discontinuation for other reason, whichever occurs first.
  Those subjects with clinical benefit from treatment (CR, PR, and SD) as per the investigator's discretion, will be allowed to continue receiving treatment with MB12/Keytruda® in the Extended Study Period, according to the arm initially assigned, every 3 weeks, for a maximum of 52 weeks from the first infusion or until evidence of disease progression, intolerance to the study drug, or treatment discontinuation for other reason, whichever occurs first.
  Interventions: Drug: Pembrolizumab
- Investigational Product (Experimental): MB12 will be administered as monotherapy, on Day 1 of every 3-week cycle (21 days), during the Main Study Period (6 cycles) unless there is disease progression, intolerance to the study drug, or treatment discontinuation for other reason, whichever occurs first.
  Those subjects with clinical benefit from treatment (CR, PR, and SD) as per the investigator's discretion, will be allowed to continue receiving treatment with MB12/Keytruda® in the Extended Study Period, according to the arm initially assigned, every 3 weeks, for a maximum of 52 weeks from the first infusion or until evidence of disease progression, intolerance to the study drug, or treatment discontinuation for other reason, whichever occurs first.
  Interventions: Drug: Pembrolizumab biosimilar

INTERVENTIONS:
Drug: Pembrolizumab — Study drug administration: intravenous infusion Dosing instructions: 200 mg administered over 30 minutes, every 3 weeks The time for infusion should be closer to 30 minutes. However, considering the variability of the infusion pumps from one center to another, a -5 to +10 minutes window is allowed (ie, the time for infusion is 30 minutes with an allowed range of 25 to 40 minutes).
  Other Names: Keytruda
  Arms: Medical Reference Product
Drug: Pembrolizumab biosimilar — Study drug administration: intravenous infusion Dosing instructions: 200 mg administered over 30 minutes, every 3 weeks The time for infusion should be closer to 30 minutes. However, considering the variability of the infusion pumps from one center to another, a -5 to +10 minutes window is allowed (ie, the time for infusion is 30 minutes with an allowed range of 25 to 40 minutes).
  Other Names: MB12
  Arms: Investigational Product

SUMMARY:
This is a randomized, multicenter, multinational, double-blind, and parallel-group study to evaluate the PK, efficacy, safety and immunogenicity of MB12 (proposed pembrolizumab biosimilar) versus Keytruda® in subjects with newly diagnosed stage IV non-squamous NSCLC. This study is planned to be conducted in approximately 48 sites in 7 countries, a total of 174 subjects will be enrolled.

Eligible subjects will be randomized in a 1:1 ratio to receive MB12 or Keytruda® at a dose of 200 mg every 3 weeks. Subjects will be stratified by gender (male versus female) and ECOG status (0 versus 1) as both factors are considered to have the potential to influence PK properties of pembrolizumab to some extent.

The study will consist of 2 periods defined as follows:

* Main Study Period from Screening up to Cycle 6 included.
* Extended Treatment Period from Cycle 7 up to Week 52 for those subjects who demonstrate clinical benefit from the treatment (complete response [CR], partial response [PR], and stable disease [SD]). They will continue treatment until disease progression, intolerance to the study drug, treatment discontinuation for other reason, or up to Week 52, whichever occurs first.

A Data Safety Monitoring Board (DSMB) will assess the safety data periodically and will recommend to the sponsor whether to continue, modify, or stop the trial on the basis of safety considerations. After the first 10 subjects have received at least 2 cycles of treatment, the DSMB will review the accumulated safety data, and the first meeting will take place. Subsequent meetings will be performed as per the DSMB charter.

DETAILED DESCRIPTION:
MB12 is being developed by mAbxience Research S.L., and its clinical development is sponsored by Laboratorio Elea Phoenix S.A. as a proposed biosimilar to Keytruda®. The reference medicinal product is European Union (EU)-sourced Keytruda®, manufactured and marketed by Merck Sharp & Dohme.

Study drugs: MB12 and Keytruda® Study drug administration: intravenous infusion Dosing instructions: 200 mg administered over 30 minutes, every 3 weeks

The study will consist of 2 periods defined as follows:

* Main Study Period from Screening up to Cycle 6 included.
* Extended Treatment Period from Cycle 7 up to Week 52 for those subjects who demonstrate clinical benefit from the treatment (CR, PR, and SD). They will continue treatment until disease progression, intolerance to the study drug, treatment discontinuation for other reason, or up to Week 52, whichever occurs first.

The anti-tumor activity will be determined by local radiological examination for all measurable and evaluable lesions according to RECIST version 1.1. During the Main Study Period, the efficacy assessments will be performed every 6 weeks from the first infusion (Cycle 1, Day 1). During the Extended Treatment Period, the assessments will be performed every 9 weeks, from Week 18 onwards, according to RECIST criteria, until disease progression, intolerance to the study drug, treatment discontinuation for other reason, or up to 52 weeks, whichever occurs first.

Safety assessments include vital signs, physical examination, ECOG performance status, 12-lead ECGs, clinical laboratory assessments (hematology, clinical chemistry, thyroid function, coagulation, virology, urinalysis, and pregnancy tests), and AE assessments.

The primary PK parameter is AUCss at Cycle 6. Serum concentrations used for estimating AUCss will be determined by a validated analytical procedure once steady state (5 elimination half-lives) has been reached.

Secondary PK parameters, including maximum concentration (Cmax), minimum concentration (Ctrough), time to maximum concentration (tmax), clearance (CL), elimination half-life (t1/2), and volume of distribution (Vss), will be calculated for Cycle 1 and Cycle 6, as applicable. Additional PK parameters may be included if deemed appropriate.

PK variables will be calculated according to the recommendations of the European Medicines Agency (EMA) and the World Health Organization (WHO).

Blood samples for PK analysis will be collected at Cycle 1 and Cycle 6 as follows: predose; at 30 minutes after the SOI; at 4, 6, 24, 48, 168, 336, and 504 hours after the SOI.

The comparison of the immunogenicity profile of MB12 versus Keytruda® during the Main Study and Extended Treatment Periods include:

* ADAs
* Nabs in ADA (+) samples
* Titers in ADA (+) samples During the Main Study Period, blood samples for immunogenicity will be collected pre-dose at Cycle 1 Day 1, Cycle 1 Day 14, pre-dose at Cycle 3 Day 1, and pre-dose at Cycle 6 Day 1. During the Extended Treatment Period, 2 additional samples will be collected in those subjects who continue treatment after Cycle 6 at Week 26 and at Week 52 or EOT/early termination (if this occurs before Week 52 and if previous sample has not been taken within the last 16 weeks).

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the following criteria to be included in the study:

1. Willing and able to provide written informed consent for the study before the initiation of any study-specific procedures.
2. Greater than or equal to 18 years of age at the time of signing the ICF.
3. Body weight ≥50 kg at Screening.
4. Having newly diagnosed stage IV (defined by the eighth edition of the TNM classification) non-squamous NSCLC, without prior systemic treatment for the disease. For those subjects in whom the pleural or pericardial effusion is the only location of metastatic disease, confirmation of its malignant etiology is required.
5. At least 1 radiographically measurable lesion per RECIST version 1.1, locally assessed.
6. Programmed death-ligand 1 (PD-L1) expression ≥50%, locally determined by immunohistochemistry, as determined by a Food and Drug Administration (FDA) validated method.
7. Life expectancy of at least 3 months.
8. ECOG performance status of 0 to 1.
9. Adequate hepatic, renal, hematologic, endocrine, and coagulation function, defined as:

   1. Liver function: bilirubin level ≤1.5 × the upper limit of normal (ULN) (≤3 × ULN for subjects with Gilbert's syndrome), albumin level ≥ lower limit of normal (LLN), aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤2.5 × ULN in subjects without liver metastases or ≤5 × ULN in subjects with liver metastases.
   2. Renal function: serum creatinine level ≤1.5 × ULN, calculated creatinine clearance ≥50 mL/min (Cockcroft-Gault formula).
   3. Hematologic function: absolute neutrophil count ≥1.5 × 109/L; platelet count ≥100 × 109/L, hemoglobin ≥9 g/dL.
   4. Endocrine function: thyroid stimulating hormone (TSH) within normal limits. If TSH is not within normal limits, the subject may still be eligible if T3 and free T4 are within normal limits.
   5. Coagulation: international normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy. Subjects on anticoagulant therapy must be on a stable anticoagulation regimen and have an INR not above the target therapeutic range for the 14 days before the first dose of the study drug.
10. Subjects with a negative COVID-19 test (done at the discretion of investigator or per local regulation) within previous 24 hours before randomization. In case of confirmed COVID-19 infection before Screening, documentation of resolution of infection by appropriate laboratory test is required.
11. No history of prior malignancy, except for basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or cervical cancer in situ, or has undergone potentially curative therapy without evidence of disease recurrence for 3 years from the start of that therapy.
12. Women of childbearing potential (WOCBP) must either abstain from sexual intercourse or employ highly effective contraception measures during the study and for at least 6 months after the last dose of the study drug. Highly effective measures include 2 forms of contraception. Postmenopausal or surgically sterile women (ie, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) are eligible. Postmenopausal status is defined as either: amenorrheic for ≥12 months following cessation of exogenous hormonal treatments and without an alternative medical cause; luteinizing hormone and follicle stimulating hormone levels in the postmenopausal range for women under 50 years of age; radiation-induced ovarian ablation with last menses ≥1 year ago; or chemotherapy-induced menopause with a ≥1-year interval since last menses. Female subjects must refrain from donating or banking eggs (ova, oocytes) and retrieving eggs for use during study treatment and for 6 months after the last dose of the study drug.
13. Male subjects, if not surgically sterile, must either abstain from sexual intercourse or employ highly effective contraception (condoms or other barrier forms of contraception) during the study and for at least 6 months after the last dose of the study drug. Male subjects should also avoid semen donation or providing semen for in-vitro fertilization during the above mentioned duration.

Exclusion Criteria:

1. Unwilling or unable to comply with scheduled visits, drug administration plan, laboratory tests, or other study procedures and study restrictions.
2. Predominantly squamous cell histology NSCLC. Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the subject is ineligible.
3. Participation in another clinical trial or treatment with another investigational agent within 4 weeks or 5 half-lives before randomization, whichever is longer.
4. Known actionable mutations for which there is an approved and available therapy.
5. Known central nervous system metastases and/or carcinomatous meningitis.
6. Previous systemic steroid therapy (prednisone at a dose of 10 mg or equivalent) within 3 days before the first dose of the study drug or receiving any other form of immunosuppressive medication. Subjects receiving daily steroid replacement therapy (daily prednisone at a dose of 5 to 7.5 mg or equivalent) could be included in the study.
7. Subject who requires any other form of localized or systemic antineoplastic therapy during the study.
8. Prior anti-programmed cell death-1 (anti-PD-1), anti-PD-L1, anti programmed death-ligand 2 (anti-PD-L2), anti-CD137, or anti cytotoxic T lymphocyte antigen (CTLA)-4 therapy (including ipilimumab or any other antibody or drug that specifically targets co stimulation of T cells or immune checkpoints).
9. Prior systemic cytotoxic chemotherapy, biological therapy, or major surgery within 3 weeks before the first dose of the study drug; have received thoracic radiation therapy of >30 gray (Gy) within 6 months before the first dose of the study drug. Palliative radiotherapy is allowed if completed >14 days before the first dose of the study drug.
10. Known history of severe hypersensitivity to another monoclonal antibody.
11. Active autoimmune disease which has required systemic treatment in the last 2 years before the first dose of the study drug (eg, disease modifying agents, corticosteroids, or immunosuppressive treatment). Replacement therapy (eg, thyroxine, insulin, or physiological corticosteroid replacement therapy for pituitary or adrenal insufficiency) is not considered a form of systemic treatment.
12. Interstitial lung disease or pneumonitis requiring oral or intravenous steroids.
13. Active infection or a previous infection requiring intravenous systemic treatment within 30 days before the first dose of the study drug.
14. Subject who has received or is about to receive a live virus vaccination within 30 days before the first dose of the study drug. Seasonal flu and COVID-19 vaccines that do not contain live virus are permitted.
15. Known history of human immunodeficiency virus (HIV)-1 or HIV-2.
16. Known active tuberculosis or hepatitis B (hepatitis B surface antigen [HBsAg] positive) or hepatitis C (hepatitis C antibody positive and hepatitis C virus [HCV] RNA positive).
17. Subject who has received a solid organ/tissue allogeneic transplant.
18. Known psychiatric disorders that could interfere with cooperation with study requirements.
19. At the time of signing the ICF, the subject is a regular user (including "recreational use") of any illicit drug or has a recent history (within the past year) of substance abuse (including alcohol).
20. Subject is pregnant or lactating or expecting to conceive during the study or up to 120 days after the last dose of the study drug.
21. Immediate family member who is at the research site or sponsoring staff who is directly involved in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
AUC (area under the curve) | Four months
  The primary PK parameter is AUC (area under the curve in the serum concentration-time plot) at Cycle 6. Serum concentrations used for estimating AUC will be determined by a validated analytical procedure once steady state (5 elimination half-lives) has been reached.
Cmax (maximum serum concentration) | Four months
  Cmax will be calculated for Cycle 1 and Cycle 6.
Tmax (time for maximum serum concentration) | Four months
  Tmax will be calculated for Cycle 1 and Cycle 6.

SECONDARY OUTCOMES:
Best overall response | 52 weeks
  To compare the best overall response (BOR) during the Main Study Period and progression-free survival (PFS) during the Extended Treatment Period of MB12 and Keytruda®.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 52 weeks
  Safety will be monitored by incidence, nature, and severity of treatment-emergent adverse events, including adverse drug reactions graded according to CTCAE version 5.0.
Number of participants developing anti-drug antibodies | 52 weeks
  Blood samples will be taken to determine ADAs through 52 weeks after the first study drug administration. Anti pembrolizumab antibodies will be presented as negative (lower than the test cut-off) or positive (above the test cut-off) and will be presented by treatment group.
  Results will be presented by summarizing frequency (n) and percentage (%) of subjects with a positive result.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Spitzer, MSc, Study Chair — Laboratorio Elea Phoenix
Locations (1):
- Clínica Viedma, Viedma, Río Negro Province, Argentina

IPD SHARING:
Plan to Share IPD: No